CLINICAL TRIAL: NCT04290078
Title: The Kaia Back Pain Intervention for Self-management of Low Back Pain - a Randomized Controlled Study
Brief Title: The Kaia Back Pain Intervention for Self-management of Low Back Pain
Acronym: BACKSPIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kaia Health Software (Industry)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KaiaBP001
Record Dates: First submitted 2020-02-18; First posted 2020-02-28 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kaia Back Pain Study Intervention (Experimental): The study intervention consists of training sessions conducted daily by the participant via Kaia back pain program. This content combines several approaches that may be effective when used together such as physical exercises, relaxation practices and learning modules. Additionally, there is availability of an electronic motion coach on a set of exercises.
  Users also receive behavioural health coaching provided by Kaia's coaching staff based on a coaching curriculum.
  Interventions: Device: Kaia Back Pain Study App
- Control Group (Active Comparator): Participants in the control arm will be provided with online links to educational materials about home exercises and pain management and asked to continue their usual care. On-line resources will include links to Web MD, the National Library of Medicine (Medline), and OnHealth.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Kaia Back Pain Study App — Kaia Back Pain is an integrated solution for self-management of low-back pain that digitizes multidisciplinary rehabilitation into a smartphone application.
  Arms: Kaia Back Pain Study Intervention
Other: Usual Care — Participants in the control arm will be provided with online links to educational materials about home exercises and pain management and asked to continue their usual care. On-line resources will include links to Web MD, the National Library of Medicine (Medline), and OnHealth
  Arms: Control Group

SUMMARY:
The study aims to evaluate outcomes of the use of Kaia Study app (software program application for self-management of low-back pain) on back pain among adults with non-specific subacute and chronic low back pain based on change in pain intensity, physical functioning, quality of life (PROMIS-10) based on self-reported information from baseline to study end as compared to a control group.

DETAILED DESCRIPTION:
This is a two-arm, parallel assignment, open-label, randomized control trial comparing back pain outcomes in an intervention group (MPT using the Kaia app) to those of a control group (usual care without restrictions on treatment). It is designed to enroll up to 184 participants. The treatment period will last for 90 days. This includes the randomization assignment and follow-up evaluations at 30 days, 60 days, and 90 days post-randomization. After pre-screening and informed consent activities are completed, the study will be conducted using electronic patient reported outcomes (ePROs); participants can complete all study tasks at home by means of internet-enabled devices. Participants assigned to the intervention group will implement Kaia's exercise regimen using their personal mobile devices. The control group will receive usual care without restrictions and will be provided with internet-based information about treatment of non-specific back pain, including handouts depicting typical home-based exercises as recommended by American Academy of Orthopedic Surgeons.

ELIGIBILITY:
Inclusion Criteria:

1. Between 22 and 75 years old
2. Able to speak, read, and understand English
3. Smartphone user with a compatible device, built-in camera, and internet access at home
4. Pain intensity ≥4/10 on Numeric Rating Scale (NRS) for low back pain, on average, in the week prior to screening
5. Low back pain diagnosis with duration ≥1 month and <12 months (i.e., non-specific subacute or chronic back pain)
6. Willingness and capable of providing Informed Consent to use the Kaia Study app and participate in all assessments associated with this clinical study

Exclusion Criteria:

1. Referral or plans for surgery, chiropractic care, acupuncture, injections or other treatment for low back pain in the next 1 month following screening
2. Self-reported prior subscription to Kaia app or plans to participate in any other investigational trials or protocols for low back pain within 90 days
3. Known pregnancy at screening or plans to become pregnant during study.
4. Prior back surgery or current workers compensation case or litigation related to back pain
5. Self-reported ongoing use of opioids for conditions other than back pain within 30 days prior to screening
6. If taking opioid or NSAID medication for back pain, changes in dosing or type of medications used for analgesic regimen within 30 days prior to screening
7. Use of opioids greater than the following daily doses: oxycodone >20 mg per day, morphine > 30 mg per day, hydrocodone > 30 mg per day, or tramadol > 300 mg per day within 30 days prior to screening
8. Self-reported history of substance abuse within 1 year
9. Diagnosis of specific underlying cause of back pain (e.g., known spinal fracture, spinal tumor, spinal infection, disc herniation, spinal stenosis)
10. Severe or unstable medical condition (e.g., unstable cardiac disease, active infection, stroke with residual neuromuscular effects, paralysis, gait imbalance, or history of recent recurrent falls)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | Change from baseline NRS at 90 days
  Pain Intensity (NRS-11, 0 no pain to 10 Severe pain)

SECONDARY OUTCOMES:
Oswestry Disability Index | baseline (day 0), day 30, day 60 and day 90
  Measure of Disability in Low Back Pain ( Scale from "0%" no disability no to "100% worst possible disability" )
Patient-Reported Outcomes Measurement Information System 10-Question Short Form (PROMIS-10) | baseline (day 0), day 30, day 60 and day 90
  Quality of Life and overall Health Status (scores are transformed to t score distributions with a mean of 50 and standard deviation of 10. A higher score indicates better health)
Perceived Treatment Helpfulness | baseline (day 0), day 30, day 60 and day 90
  Feedback on the mobile medical application (5-Point Likert Scales ranging from 1 "lowest satisfaction" to 5 "highest satisfaction")
Pain Catastrophizing Scale | baseline (day 0) and at day 90
  Quantify individual's pain catastrophizing (scored from 0 "no catastrophizing" to 52 "worst possible catastrophizing")
Satisfaction and perceived treatment helpfulness | Study End at day 90
  Feedback on the mobile medical application (5-Point Likert Scales ranging from 1 "lowest satisfaction" to 5 "highest satisfaction")
Health care utilisation | baseline (day 0), day 30, day 60 and day 90
  Use of services by persons for the purpose of preventing and curing health problems (type and number of times utilized)
Change in concomitant medication use | baseline (day 0), day 15, day 30, day 45, day 60, day 75 and day 90
  Record of intaken concomitant analgetic medication (number of uses)
Number of Adverse Events | baseline (day 0), day 15, day 30, day 45, day 60, day 75 and day 90
  Absolute number of untoward medical occurrences
Number of Device Deficiencies | baseline (day 0), day 15, day 30, day 45, day 60, day 75 and day 90
  Absolute number of untoward technical occurrences

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Srdjan Nedeljkovic, MD, Principal Investigator — Physiatry, Spine & Pain Management
Locations (1):
- Brigham and Women's Hospital /Physiatry, Spine & Pain Management, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No